CLINICAL TRIAL: NCT05769296
Title: Australian UCSF Concussion in Athletes Studied With Cranial Accelerometry
Brief Title: Australian UCSF Concussion in Athletes
Acronym: AUSSIE-1
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 1572
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Concussion, Mild
Keywords: mild traumatic brain injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concussed: Diagnosis of concussion
  Interventions: Device: Headpulse measurements
- Controls: Athletes with no concussion within the preceding year
  Interventions: Device: Headpulse measurements

INTERVENTIONS:
Device: Headpulse measurements — Placement of headset on subject

SUMMARY:
Analysis of cardiac induced brain forces using cranial accelerometry has been shown to diagnose concussion in high school athletes. This trial expands on this observation by recording headpulse signals in a recently concussed athletes playing Australian rules football.

DETAILED DESCRIPTION:
Recently concussed athletes will have headpulse measurements obtained as soon after the clinically identified concussion as is feasible and at 1-3 day intervals over the course of a month. These recordings will pair with a self administered neurological symptom inventory (NSI) to track the athletes subjective concussion symptoms. Data will be used to confirm prior models of analysis and produce a tool to be confirmed in a future study.

ELIGIBILITY:
Concussion Subjects:

Inclusion Criteria:

* Diagnosed with sport related concussion
* first recording obtained within one week
* willingness to have multiple recordings in the month following concussion

Exclusions:

- head laceration

Control subjects:

Inclusion Criteria:

* athletes without concussion over the last year
* willingness to have single or multiple recordings

Exclusion Criteria:

- head laceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recently concussed athletes playing Australian rules football. Controls are athletes of Australian Football or other sports without concussion for more than 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of headpulse measurements to detect subjects with concussion | 1 month
  Proportion of clinically concussed athletes that have headpulse values > 2SD of control subjects

SECONDARY OUTCOMES:
Feasibility of subject recruitment | 2.5 months
  Number of subjects recruited during playoff season

CONTACTS AND LOCATIONS:
Overall Officials: Wade S Smith, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No